CLINICAL TRIAL: NCT06274775
Title: Effect of an Educational Nail Biopsy Video on Pre-operative Anxiety, Health Literacy, and Patient Satisfaction: a Single Center Randomized Controlled Trial
Brief Title: Effect of an Educational Nail Biopsy Video on Pre-operative Anxiety, Health Literacy, and Patient Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 23-12026811
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Literacy; Satisfaction, Patient
MeSH Terms: conditions — Anxiety Disorders; Literacy; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video Group (Experimental): Group A (intervention group), which will be shown an educational video about the nail biopsy procedure in addition to standard of care, which includes verbal information about the procedure and pre-operative and post-operative handouts with instructions provided via quick-response (QR) code.
  Interventions: Other: Educational Video
- Standard of Care Group (No Intervention): Standard of care only, which includes verbal information about the procedure and pre-operative and post-operative handouts with instructions provided via quick-response (QR) code.

INTERVENTIONS:
Other: Educational Video — Educational video about the nail biopsy procedure
  Arms: Educational Video Group

SUMMARY:
The investigators are interested in studying the effect of an animated video depicting a nail biopsy procedure on the anxiety, health literacy, and satisfaction of participants recommended to undergo a nail biopsy procedure. The investigators hypothesize that the animated video will reduce preoperative anxiety, increase health literacy, and increase patient satisfaction in relation to nail biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients recommended to receive a nail biopsy procedure in our specialty nail clinic.

Exclusion Criteria:

* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety, as measured by the State Trait Anxiety Inventory | Immediately following nail biopsy consultation
  State Trait Anxiety Inventory uses a scale of 1-4 for each question, with 1 being "not at all" and 4 being "very much so." The maximum score is 80, and the minimum score is 20. Scores from 20-37 indicate "no or low anxiety," scores from 38-44 indicate "moderate anxiety," and scores from 45-80 indicate "high anxiety."
Anxiety, as measured by the Amsterdam Preoperative Anxiety and Information Scale | Immediately following nail biopsy consultation
  The Amsterdam Preoperative Anxiety and Information Scale uses a Likert scale from 1-5. The questions focus on anxiety and the need for information, creating two separate sub-scores. This measure assesses the anxiety sub-score, which ranges from 4 to 20 (4 questions) A higher anxiety sub-score indicates a higher anxiety level.
Need for information, as measured by the Amsterdam Preoperative Anxiety and Information Scale | Immediately following nail biopsy consultation
  The Amsterdam Preoperative Anxiety and Information Scale uses a Likert scale from 1-5. The questions focus on anxiety and the need for information, creating two separate sub-scores. This measure assesses the need for information sub-score, which ranges from 2 to 10 (2 questions). A higher need for information sub-score indicates a higher information requirement.
Health literacy, as measured by 4 domains of The Health Literacy Questionnaire | Immediately following nail biopsy consultation
  Using 4 domains of the The Health Literacy Questionnaire, subjects will respond using a scale from "strongly disagree" (equivalent to 1 point on Likert scale) to "strongly agree" (equivalent to 4 points on Likert scale) or from "cannot do or always difficult" (equivalent to 1 point on Likert scale) to "always easy" (equivalent to 5 points on Likert scale). The maximum score is 86, the minimum score is 19. A higher score indicates higher health literacy, while a lower score indicates lower health literacy.
Patient satisfaction, as measured by a patient satisfaction survey | Immediately following nail biopsy consultation
  The patient satisfaction survey uses a scale from "not at all" (equivalent to 1 on a Likert scale) to "very much" (equivalent to 4 on a Likert scale), or from "not acceptable" (equivalent to 1 on a Likert scale) to "Acceptable" (equivalent to 3 on a Likert scale). The maximum score is 27, the minimum score is 7, with a higher score indicating higher satisfaction, and a lower score indicating lower satisfaction.

SECONDARY OUTCOMES:
Quality of video intervention for intervention participants, as measured by a qualitative feedback survey | Immediately following nail biopsy consultation
  The qualitative survey focuses on themes of interest, understandability, video length, and whether 2D animation is an effective method to convey medical information.

CONTACTS AND LOCATIONS:
Overall Officials: Shari R. Lipner, MD, PhD, Principal Investigator — Weill Cornell Medicine, Department of Dermatology
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DK, Chang MJ, Desai AD, Lipner SR. Clinical and dermoscopic findings of benign longitudinal melanonychia due to melanocytic activation differ by skin type and predict likelihood of nail matrix biopsy. J Am Acad Dermatol. 2022 Oct;87(4):792-799. doi: 10.1016/j.jaad.2022.06.1165. Epub 2022 Jun 22. PMID 35752275
- [Background] Turkdogan S, Roy CF, Chartier G, Payne R, Mlynarek A, Forest VI, Hier M. Effect of Perioperative Patient Education via Animated Videos in Patients Undergoing Head and Neck Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Feb 1;148(2):173-179. doi: 10.1001/jamaoto.2021.3765. PMID 34967863
- [Background] Hou H, Li X, Song Y, Ji Y, Sun M, Wang D, Jiao J, Qu J, Gu H. Effect of interactive, multimedia-based home-initiated education on preoperative anxiety inchildren and their parents: a single-center randomized controlled trial. BMC Anesthesiol. 2023 Mar 28;23(1):95. doi: 10.1186/s12871-023-02055-7. PMID 36977985